CLINICAL TRIAL: NCT05706844
Title: Randomized Trial on Spinal Anaesthesia vs. General Anaesthesia (SAGA) on Recovery After Total Hip, Total Knee, and Unicompartmental Knee Arthroplasty
Brief Title: Spinal Anaesthesia vs. General Anaesthesia for THA, TKA and UKA
Acronym: RCT SAGA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anders Troelsen (Other)
Collaborators: Vejle Hospital (Other)
Responsible Party: Sponsor-Investigator, Anders Troelsen, Professor, consultant physician, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-501221-21-00
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: Hip arthroplasty; Knee arthroplasty; Unicompartmental knee arthroplasty; General anaesthesia; Spinal anaesthesia; Hip osteoarthritis; Knee osteoarthritis; Fast-track surger
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Each of the three arthroplasty procedures are investigated in a 2-arm randomised trial:
  Total hip arthroplasty - either spinal anaesthesia or general anaesthesia.
  Total knee arthroplasty - either spinal anaesthesia or general anaesthesia.
  Unicompartmental knee arthroplasty - either spinal anaesthesia or general anaesthesia.
Who Masked: Outcomes Assessor
Masking Description: Physcians and nurses in the surgical department are not able to be blinded. But outcome assesors (ie. physiotherapists, research personel) are not aware of the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal Anaesthesia (SA) (Experimental): Patients undergoing total hip, total knee or unicompartmental knee arthroplasty are anaesthetized using:
  Plain or heavy Bupivacaine hydrochloride 10 mg (2 mL)
  Interventions: Drug: Spinal anesthesia
- General Anaesthesia (GA) (Experimental): Patients undergoing total hip, total knee or unicompartmental knee arthroplasty are anaesthetized using:
  Propofol (induction: 1.0-2.0 mg/kg. infusion: 3-5 mg/kg/hour) + Remifentanil (induction: 3-5 mcg/kg, infusion: 0.5 mcg/kg/min)
  Interventions: Drug: General anaesthesia

INTERVENTIONS:
Drug: Spinal anesthesia — plain or heavy Bupivacaine hydrochloride 10 mg (2 mL) injected in the spinal canal
  Other Names: Spinal anaesthesia
  Arms: Spinal Anaesthesia (SA)
Drug: General anaesthesia — Propofol (induction: 1.0-2.0 mg/kg. infusion: 3-5 mg/kg/hour) + Remifentanil (induction: 3-5 mcg/kg, infusion: 0.5 mcg/kg/min) given intravenously
  Arms: General Anaesthesia (GA)

SUMMARY:
The goal of this randomized clinical trial is to investigate the postoperative recovery following hip and knee arthroplasty procedures depending on the use of either spinal anaesthesia (SA) or general anaesthesia (GA).

The main questions are:

* Are more patients able to be safely mobilized within 6 hours postoperatively when using GA compared to SA?
* Does postoperative pain, nausea and vomiting, dizzyness, occurence of delirium and urinary retention differ between the anaesthetic methods?

Participants, scheduled for total hip, total knee and unicomartmental knee arthroplasty, will be randomized to recieve spinal anaesthesia or general anaesthesia in relation to surgery. At 6 hours postoperatively a physiotherapist will conduct a 5-meter walking test to evaluate whether the participant can be safely mobilized.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological hip or knee osteoarthritis meeting the indications for primary total hip, total knee, or unicompartmental knee arthroplasty.
* ≥18 years of age.
* Able to speak and understand Danish
* Able to give informed consent and must be cognitively intact.

Exclusion Criteria:

* Lives in an institution.
* Uses walking aid such as a walker or a wheelchair.
* Terminal illness.
* Has contraindications for either general or spinal anaesthesia.
* Has objections to receiving either general or spinal anaesthesia.
* Requires anxiolytics as premedication prior to anaesthesia.
* Traumatic aetiology as a basis for surgical indication.
* Altered pain perception and / or neurologic affection due to diabetes or other disorders.
* Daily preoperative use of opioids > 30 mg of morphine milligram equivalents (MME).
* Standard primary arthroplasty procedure is evaluated not to be suitable.
* Women considered fertile but without sufficient birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Ability to be mobilsed safely within 6 hours of surgery | within 6 hours postoperatively.
  5-meter walking test where a physiotherapist evaluates whether the participant can be safely mobilized within 6 hours of surgery.

SECONDARY OUTCOMES:
Fulfilment of discharge criteria | On the day of surgery: at 4 hours postoperatively and 6 hours postoperatively. From postoperative day 1 and until discharge (on average 1 day): at 10.00 and at 18.00. This will be asses as long as the patient is admitted.
  Dichotomous (Yes or No)
Pain score | On the day of surgery: at 4 hours postoperatively and 6 hours postoperatively. From postoperative day 1 and until discharge (on average 1 day): at 10.00 and at 18.00. This will be asses as long as the patient is admitted.
  Will be recorded during rest and 5-m walk using participant evaluated NRS of 0 to 10, with 10 being worst pain/dizziness/nausea imaginable. This will be recorded at 4 and 6 hours post-operatively on the day of surgery and at 10:00 and 18:00 on the following postoperative days.
Opioid use in Morphine Milligram Equivilents within the first 6 hours of surgery | On the day of surgery: Within the first 6 hours after surgery.
  Cumulated opioid use in Morphine Milligram Equivalents.
Nausea Score | On the day of surgery: at 4 hours postoperatively and 6 hours postoperatively. From postoperative day 1 and until discharge (on average 1 day): at 10.00 and at 18.00. This will be asses as long as the patient is admitted.
  Will be recorded during rest and 5-m walk using participant evaluated NRS of 0 to 10, with 10 being worst pain/dizziness/nausea imaginable. This will be recorded at 4 and 6 hours post-operatively on the day of surgery and at 10:00 and 18:00 on the following postoperative days.

OTHER OUTCOMES:
Vital signs - systolic blood pressure | On the day of surgery: at 4 hours postoperatively and 6 hours postoperatively. From postoperative day 1 and until discharge (on average 1 day): at 10.00 and at 18.00. This will be asses as long as the patient is admitted.
  Systolic blood pressure (mmHg).
Vital signs - diastolic blood pressure | On the day of surgery: at 4 hours postoperatively and 6 hours postoperatively. From postoperative day 1 and until discharge (on average 1 day): at 10.00 and at 18.00. This will be asses as long as the patient is admitted.
  Diastolic blood pressure (mmHg).
Quality of Recovery-15 score | On the day of surgery: at 4 hours postoperatively. From postoperative day 1 and until discharge (on average 1 day): at 10.00. This will be asses as long as the patient is admitted.
  Four hours postoperatively on the day of surgery and at 10:00 on the following

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, MD, DMSc, Principal Investigator — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Christian Bredgaard Jensen, Hvidovre
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT05706844/SAP_000.pdf